CLINICAL TRIAL: NCT01359410
Title: Effect of a Reinforced Staple Line on Leak Rate in Distal Pancreatectomy
Brief Title: Reinforced Staple Line on Leak Rate in Distal Pancreatectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The 3rd interim analysis found superiority in the mesh reinforcement arm
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-1192
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreas adenocarcinoma; Precancerous lesions of the pancreas (mucinous cystic neoplasms, IPMN); Pancreas neuroendocrine cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant's were blinded to the results of the randomization for 6 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stapled transection with mesh reinforcement (Active Comparator): Mesh reinforced staple line (SEAMGUARD® or PERI-STRIPS DRY®)
  Interventions: Device: Mesh reinforced staple line (SEAMGUARD); Device: Stapled without mesh reinforcement (PER-STRIPS DRY)
- Stapled transection without mesh reinforcement (No Intervention)

INTERVENTIONS:
Device: Mesh reinforced staple line (SEAMGUARD) — Reinforce the pancreatic transaction with SEAMGUARD®
  Arms: Stapled transection with mesh reinforcement
Device: Stapled without mesh reinforcement (PER-STRIPS DRY) — Stapled without mesh reinforcement (PERI-STRIPS DRY®)
  Arms: Stapled transection with mesh reinforcement

SUMMARY:
The investigators propose a randomized, controlled trial of stapled pancreatic transection versus mesh reinforced stapled pancreatic transection. For the duration of the study period, participating surgeons will utilize a standardized staple technique. Either a reabsorbable polytrimethylene carbonate mesh (SEAMGUARD®) or reabsorbable strips of bovine pericardium (PERI-STRIPS DRY®) will be used to reinforce the stapled pancreatic transection line in the test group. In order to have a uniform test method, the investigators will utilize a laparoscopic stapling device for both open and laparoscopic procedures and a uniform staple size (4.8mm).

DETAILED DESCRIPTION:
Pancreatic leak remains a significant cause of morbidity and extra cost following distal pancreatectomy. Historically, previous attempts to reduce the leak rate have met with limited success. To examine this problem the investigators propose a randomized, controlled trial of stapled pancreatic transection versus mesh reinforced stapled pancreatic transection. For the duration of the study period, participating surgeons will utilize a standardized staple technique. Either a reabsorbable polytrimethylene carbonate mesh (SEAMGUARD®) or reabsorbable strips of bovine pericardium (PERI-STRIPS DRY®) will be used to reinforce the stapled pancreatic transection line in the test group. In order to have a uniform test method, the investigators will utilize a laparoscopic stapling device for both open and laparoscopic procedures and a uniform staple size (4.8mm). A drain will be placed in the left upper quadrant at the time of resection. Drainage of the pancreatic resection bed is widely accepted and remains our current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older and able to give consent. Any patient undergoing a distal pancreatectomy, laparoscopic or open, will be eligible for randomization.
* No exclusion is provided for primary diagnosis. In the event of a patient undergoing a planned resection of another organ or organs with only a possibility of a distal pancreatic resection (i.e. colectomy, hepatectomy, gastrectomy, nephrectomy), the patient will still be eligible for inclusion in the study. We expect that some patients will be randomized but not resected (ie metastasis identified). A few patients may not be stapled using the study device for technical reasons (ie the stapler does not fit). The data will be analyzed in an intent-to-treatment approach.

Exclusion Criteria: None specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Hawkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hawkins WG. To mesh or not to mesh, that is the question: comment on "Use of Seamguard to prevent pancreatic leak following distal pancreatectomy". Arch Surg. 2009 Oct;144(10):899. doi: 10.1001/archsurg.2009.34. No abstract available. PMID 19852096
- [Background] Johnston FM, Cavataio A, Strasberg SM, Hamilton NA, Simon PO Jr, Trinkaus K, Doyle MB, Mathews BD, Porembka MR, Linehan DC, Hawkins WG. The effect of mesh reinforcement of a stapled transection line on the rate of pancreatic occlusion failure after distal pancreatectomy: review of a single institution's experience. HPB (Oxford). 2009 Feb;11(1):25-31. doi: 10.1111/j.1477-2574.2008.00001.x. PMID 19590620
- [Background] Thaker RI, Matthews BD, Linehan DC, Strasberg SM, Eagon JC, Hawkins WG. Absorbable mesh reinforcement of a stapled pancreatic transection line reduces the leak rate with distal pancreatectomy. J Gastrointest Surg. 2007 Jan;11(1):59-65. doi: 10.1007/s11605-006-0042-6. PMID 17390188
- [Derived] Hamilton NA, Porembka MR, Johnston FM, Gao F, Strasberg SM, Linehan DC, Hawkins WG. Mesh reinforcement of pancreatic transection decreases incidence of pancreatic occlusion failure for left pancreatectomy: a single-blinded, randomized controlled trial. Ann Surg. 2012 Jun;255(6):1037-42. doi: 10.1097/SLA.0b013e31825659ef. PMID 22534422
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 06/28/2007 and closed to participant enrollment on 10/28/2011.
Pre-assignment Details: 112 participants were enrolled to the study but 12 participants (1 participant declined to be in the study and 11 participants were found to be ineligible) were excluded from the study before randomization to the arms.
Period: Overall Study
Arm/Group | Stapled Transection With Mesh Reinforcement | Stapled Transection Without Mesh Reinforcement
Started | 54 | 46
Completed | 54 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stapled Transection With Mesh Reinforcement | Stapled Transection Without Mesh Reinforcement | Total
Number analyzed (Participants) | 54 | 46 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (15.6) | 58.6 (13.4) | 58.0 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 21 | 55
  Male | 20 | 25 | 45
Region of Enrollment [Number; unit: participants]
  United States | 54 | 46 | 100
Indication for operation [Count of Participants; unit: Participants]
  Adenocarcinoma | 8 | 10 | 18
  Neuroendocrine tumor | 12 | 14 | 26
  Metastatic tumor to pancreas | 3 | 3 | 6
  Benign pancreatic tumor | 24 | 13 | 37
  Chronic pancreatitis | 3 | 4 | 7
  Normal pancreas | 4 | 2 | 6
Smoking history [Count of Participants; unit: Participants]
  Nonsmoker | 34 | 26 | 60
  Smoker | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Postoperative Pancreatic Leak at Any Time as Defined by the ISGPF Pancreatic Leak Grading System
Description: * Identified as being a grade B or grade C fistula or any fistula that altered the patients' management in any way
  * Determination of severity of pancreatic fistula was done using the ISGPF(International Study Group Pancreatic Fistula) leak/fistula/pancreatic occlusion failure
  * Grade B: >3x normal serum amylase, often well clinical condition, yes/no specific treatment, negative/positive ultrasound/CT, usually persistent drainage (>3 weeks), yes/no signs of infection, yes/no readmission, no sepsis, no reoperation, no death related to fistula
  * Grade C: >3x normal serum amylase, ill appearing/bad, requires specific treatment, positive ultrasound/CT, persistent drainage (>3 weeks), signs of infection, yes/no readmission, sepsis, reoperation, and death related to fistula
Time Frame: 100 days or removal of drain
Population: (1) participant in the mesh reinforcement arm was not evaluable due to death and (1) participant in the non-mesh reinforcement arm was not evaluable due to death.
Measure: Count of Participants; unit: Participants
Arm/Group | Stapled Transection With Mesh Reinforcement | Stapled Transection Without Mesh Reinforcement
Number analyzed (Participants) | 53 | 45
Participants | 1 | 11

2. Secondary Outcome: Occurrence of Any Fistula as Defined by the ISGPF Pancreatic Leak Grading System
Time Frame: 100 days or removal of drain
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stapled Transection With Mesh Reinforcement | Stapled Transection Without Mesh Reinforcement
Number analyzed (Participants) | 53 | 45
Participants | 21 | 26

3. Secondary Outcome: Time to Drain Removal
Time Frame: 100 days or removal of drain
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Stapled Transection With Mesh Reinforcement | Stapled Transection Without Mesh Reinforcement
Number analyzed (Participants) | 53 | 45
days | 9 [6 to 19] | 17 [7 to 40]

4. Secondary Outcome: Number of Non-pancreatic Adverse Events
Time Frame: 100 days or removal of drain
Measure: Number; unit: non-pancreatic adverse events
Arm/Group | Stapled Transection With Mesh Reinforcement | Stapled Transection Without Mesh Reinforcement
Number analyzed (Participants) | 54 | 46
non-pancreatic adverse events | 21 | 28

5. Post Hoc Outcome: Intraoperative Complications Incurred by Participants
Time Frame: 100 days or removal of drain
Measure: Number; unit: intraoperative complications
Arm/Group | Stapled Transection With Mesh Reinforcement | Stapled Transection Without Mesh Reinforcement
Number analyzed (Participants) | 54 | 46
intraoperative complications
  Staple misfire splenic artery requiring revision | 0 | 1
  Bleeding at staple line | 0 | 1
  Hepatic artery injury | 1 | 0
  Umbilical tape in staple line requiring revision | 2 | 0
  Pulmonary embolus | 1 | 0
  Splenic avulsion | 1 | 0
  Deserosalization of stomach | 1 | 0

ADVERSE EVENTS:
Arm/Group | Stapled Transection With Mesh Reinforcement | Stapled Transection Without Mesh Reinforcement
Serious Adverse Events (participants affected / at risk) | 1/54 | 11/46
Other Adverse Events (participants affected / at risk) | 3/54 | 5/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stapled Transection With Mesh Reinforcement (N=54) | Stapled Transection Without Mesh Reinforcement (N=46)
Fistula (leak) (Gastrointestinal disorders) | 1 | 11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stapled Transection With Mesh Reinforcement (N=54) | Stapled Transection Without Mesh Reinforcement (N=46)
Cerebrovascular accident (Vascular disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postoperative bleeding requiring transfusion (General disorders) | 0 | 1
Postoperative bleeding requiring reoperation (General disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute renal failure (not requiring dialysis) (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
New onset diabetes (Metabolism and nutrition disorders) | 0 | 1
Gastrointestinal bleed (Gastrointestinal disorders) | 0 | 1
Gastrointestinal anastomosis leak (Gastrointestinal disorders) | 1 | 1
Prolonged ileus (Gastrointestinal disorders) | 2 | 2
Other intraabdominal abscess (Gastrointestinal disorders) | 1 | 2
Anaphylactic reaction to medication (Immune system disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vascular psedoaneurysm (Vascular disorders) | 0 | 2
IV infiltration with skin necrosis (Injury, poisoning and procedural complications) | 1 | 0
Wound infection (Injury, poisoning and procedural complications) | 2 | 5

LIMITATIONS AND CAVEATS:
The investigators were unable to identify any complications directly due to the mesh materials. It is possible these complications are very rare and that the study did not include enough participants to potentially identify these potential harms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes